CLINICAL TRIAL: NCT01850979
Title: Treatment of Dry Eye Using 0.03% Tacrolimus Eye Drops: Prospective Double-Blind Randomized Study
Brief Title: Treatment of Dry Eye Using 0.03% Tacrolimus Eye Drops
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Fernando Eiji Sakassegawa Naves, physician, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1307/09
Record Dates: First submitted 2013-05-01; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Sjogren Syndrome; Dry Eye Syndrome
Keywords: CYCLOSPORINE/TACROLIMUS [VA Drug Interaction]
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes | interventions — Tacrolimus; Olive Oil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tacrolimus (Active Comparator): tacrolimus 0,03% eye drops (olive oil as vehicle) every 12/12 hours for 3 months placebo as olive oil eye drops every 12/12h hours for 3 months
  Interventions: Drug: Tacrolimus
- Olive Oil (Placebo Comparator): All patients in this groups receive eye drops containing olive oil (vehicle of tacrolimus eye drops) twice a day (every 12 hours) for 90 days.
  Interventions: Drug: Olive Oil

INTERVENTIONS:
Drug: Tacrolimus — tacrolimus 0,03% eyedrops (olive oil vehicle) every 12 hours for 3 months placebo : olive oil eyedrops every 12 hours for 3 months
  Other Names: FK 506
  Arms: tacrolimus
Drug: Olive Oil — All patients in this groups receive eye drops containing olive oil (vehicle of tacrolimus eye drops) twice a day (every 12 hours) for 90 days.
  Other Names: placebo
  Arms: Olive Oil

SUMMARY:
Aqueous deficiency dry eye is mainly caused by Sjogren syndrome (SS), an autoimmune, chronic, inflammatory and systemic disease which affects most commonly the lacrimal and salivary glands.The ocular treatment is focused in increasing lubrification and decreasing inflammation with topical autologous serum, topical immunosuppressive agents and corticotherapy. Use of topical immunosuppressants has increased in recent years because the topical corticotherapy leads to ocular complications. The most used immunosuppressant is cyclosporine. Tacrolimus , another immunosuppressant, has been used in treatment of immune and inflammatory ocular diseases.This study describes a prospective controlled double-blinded randomized study of the clinical outcome of SS dry eyes patients treated with 0.03% tacrolimus eye drops. As secondary purposes, outcome of dry eye symptoms and any ocular symptoms of the eye drops were also questioned to the patients.

DETAILED DESCRIPTION:
Aqueous deficiency dry eye is mainly caused by Sjogren syndrome (SS), an autoimmune, chronic, inflammatory and systemic disease which affects most commonly the lacrimal and salivary glands. The hyperreactivity of B lymphocytes causes lymphoplasmacytic infiltration, which induces production of antibodies against antigens of the acinar epithelium and ducts of the lacrimal exocrine gland . The ocular treatment is focused in increasing lubrification and decreasing inflammation with topical autologous serum, topical immunosuppressive agents and corticotherapy. Use of topical immunosuppressants has increased in recent years because the topical corticotherapy leads to ocular complications.

Among topical immunosuppressants the most used ones are tacrolimus, also known as FK506 and cyclosporine A (CsA). Their mechanism of action is similar, but FK 506 is described to be 10 to 100 times more potent than CsA. Tacrolimus is a macrolide with immunomodulatory action and becomes biologically active only when it binds to immunophilin and acts by inhibiting calcineurin, limiting transduction of the signal that carries information from the cell membrane to the nucleus, with the aim of stimulating interleukin (IL) - 2 synthesis, and inhibiting T and B lymphocyte activation . Generally, tacrolimus suppresses the immune response by inhibiting the release of other inflammatory cytokines (eg, IL-3, IL-4, IL-5, IL-8, interferon- ϒ, and tumor necrosis factor - α) .

The systemic and topical use of tacrolimus is already well established in ophthalmologic treatments of immune-mediated diseases , uveitis, graft-versus-host disease , corneal transplants and ocular pemphigoid . In veterinary medicine, topical tacrolimus aqueous suspension is well established to treat dry eye in dogs . In humans, tacrolimus eye drops were reported to be effective in treating severe allergic conjunctivitis . In a previous report, our group has showed the clinical outcomes of a case series of eight patients with dry eye using 0.03% tacrolimus eye drops 5 based on evidence in treating animals with KCS.

This study describes a prospective controlled double-blinded randomized study of the clinical outcome of SS dry eyes patients treated with 0.03% tacrolimus eye drops. As secondary purposes, outcome of dry eye symptoms and any ocular symptoms of the eye drops were also questioned to the patients.

ELIGIBILITY:
Inclusion Criteria:

* SS was diagnosed according to the SS European Criteria
* chronic symptoms of burning, foreign body sensation, itching in both eyes
* daily need of artificial tears
* abnormal Schirmer (ST) I test < 5mm or rose Bengal staining (RBS) ≥ 4, or break up time (BUT) < 5 seconds.

Exclusion Criteria:

* any structural abnormalities (lid scarring, entropion, trichiasis, etc.)
* any inflammation or active structural change in the iris or anterior chamber
* glaucoma
* previous eye surgery or punctual occlusion
* use of any other topical medication other than artificial tears
* any systemic or topical antibacterial or antiinflammatory drug treatment 90 days before study entry
* contact lens wearer
* the presence of any corneal infection
* any corneal diseases (marginal ulcer, opacity, scar, bullous keratopathy, conjunctivochalasis, symblepharon or tumor)
* pregnancy
* change in the immunosuppressive systemic therapy 90 days before study entry

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quantity of lacrimal film | 90 days
  Schirmer I test was performed using a Whatman 41 paper strip placed in the lateral lower conjunctival sac, and the measurement was recorded after 5 minutes (at least 30 minutes after BUT and staining scoring).The exam was made in the same room with control of humidity and temperature by the same examinator

SECONDARY OUTCOMES:
Evaluation of quality of lacrimal film | 90 days
  The BUT(break up time) was measured 3 times and averaged, using a chronometer in the same room with control of temperature and humidity by the same examinator.

OTHER OUTCOMES:
Evaluation of ocular surface | 90 days
  The rose bengal and fluorescein scores were performed by instilling 3 µL of a preservative-free combination of 1% rose Bengal and 1% fluorescein into the conjunctival sac according to the double vital staining method. The BUT was measured 3 times and averaged. The ocular surface staining score was rated from 0-3 (0= no staining, 1 = mild staining, 2 = moderated staining and 3 = extensive staining) . The exam was made in the same room with control of humidity and temperature by the same examinator

CONTACTS AND LOCATIONS:
Overall Officials: ruth m santo, assistent, Study Chair — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Felberg S, Dantas PE. [Sjogren's syndrome: diagnosis and treatment]. Arq Bras Oftalmol. 2006 Nov-Dec;69(6):959-63. doi: 10.1590/s0004-27492006000600032. Portuguese. PMID 17273698
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Management and therapy of dry eye disease: report of the Management and Therapy Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):163-78. doi: 10.1016/s1542-0124(12)70085-x. PMID 17508120
- [Background] Shoji J, Sakimoto T, Muromoto K, Inada N, Sawa M, Ra C. Comparison of topical dexamethasone and topical FK506 treatment for the experimental allergic conjunctivitis model in BALB/c mice. Jpn J Ophthalmol. 2005 May-Jun;49(3):205-10. doi: 10.1007/s10384-004-0187-3. PMID 15944824
- [Background] Moscovici BK, Holzchuh R, Chiacchio BB, Santo RM, Shimazaki J, Hida RY. Clinical treatment of dry eye using 0.03% tacrolimus eye drops. Cornea. 2012 Aug;31(8):945-9. doi: 10.1097/ICO.0b013e31823f8c9b. PMID 22511024
- [Background] Attas-Fox L, Barkana Y, Iskhakov V, Rayvich S, Gerber Y, Morad Y, Avni I, Zadok D. Topical tacrolimus 0.03% ointment for intractable allergic conjunctivitis: an open-label pilot study. Curr Eye Res. 2008 Jul;33(7):545-9. doi: 10.1080/02713680802149115. PMID 18600486
- [Background] Bertelmann E, Pleyer U. Immunomodulatory therapy in ophthalmology - is there a place for topical application? Ophthalmologica. 2004 Nov-Dec;218(6):359-67. doi: 10.1159/000080937. PMID 15564752
- [Background] Fei WL, Chen JQ, Yuan J, Quan DP, Zhou SY. Preliminary study of the effect of FK506 nanospheric-suspension eye drops on rejection of penetrating keratoplasty. J Ocul Pharmacol Ther. 2008 Apr;24(2):235-44. doi: 10.1089/jop.2007.0059. PMID 18321198
- [Background] Fujita E, Teramura Y, Mitsugi K, Ninomiya S, Iwatsubo T, Kawamura A, Kamimura H. Absorption, distribution, and excretion of 14C-labeled tacrolimus (FK506) after a single or repeated ocular instillation in rabbits. J Ocul Pharmacol Ther. 2008 Jun;24(3):333-43. doi: 10.1089/jop.2007.0086. PMID 18476802
- [Background] Fujita E, Teramura Y, Shiraga T, Yoshioka S, Iwatsubo T, Kawamura A, Kamimura H. Pharmacokinetics and tissue distribution of tacrolimus (FK506) after a single or repeated ocular instillation in rabbits. J Ocul Pharmacol Ther. 2008 Jun;24(3):309-19. doi: 10.1089/jop.2007.0083. PMID 18476801
- [Background] Pleyer U, Lutz S, Jusko WJ, Nguyen KD, Narawane M, Ruckert D, Mondino BJ, Lee VH, Nguyen K. Ocular absorption of topically applied FK506 from liposomal and oil formulations in the rabbit eye. Invest Ophthalmol Vis Sci. 1993 Aug;34(9):2737-42. PMID 7688360
- [Background] Ohashi Y, Ebihara N, Fujishima H, Fukushima A, Kumagai N, Nakagawa Y, Namba K, Okamoto S, Shoji J, Takamura E, Hayashi K. A randomized, placebo-controlled clinical trial of tacrolimus ophthalmic suspension 0.1% in severe allergic conjunctivitis. J Ocul Pharmacol Ther. 2010 Apr;26(2):165-74. doi: 10.1089/jop.2009.0087. PMID 20307214
- [Background] Dhaliwal JS, Mason BF, Kaufman SC. Long-term use of topical tacrolimus (FK506) in high-risk penetrating keratoplasty. Cornea. 2008 May;27(4):488-93. doi: 10.1097/ICO.0b013e3181606086. PMID 18434855
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] van Bijsterveld OP. Diagnostic tests in the Sicca syndrome. Arch Ophthalmol. 1969 Jul;82(1):10-4. doi: 10.1001/archopht.1969.00990020012003. No abstract available. PMID 4183019
- [Background] Toda I, Tsubota K. Practical double vital staining for ocular surface evaluation. Cornea. 1993 Jul;12(4):366-7. doi: 10.1097/00003226-199307000-00015. No abstract available. PMID 7687944
- [Derived] Moscovici BK, Holzchuh R, Sakassegawa-Naves FE, Hoshino-Ruiz DR, Albers MB, Santo RM, Hida RY. Treatment of Sjogren's syndrome dry eye using 0.03% tacrolimus eye drop: Prospective double-blind randomized study. Cont Lens Anterior Eye. 2015 Oct;38(5):373-8. doi: 10.1016/j.clae.2015.04.004. Epub 2015 May 5. PMID 25956572